CLINICAL TRIAL: NCT02411812
Title: Effects of the Herbst Appliance With Skeletal Anchorage or Dental Anchorage, and Twin-Block Appliance in Class II Malocclusion: A Randomized Clinical Trial
Brief Title: Effects of the Herbst Appliance With Different Anchorages and Twin-Block Appliance in Class II Malocclusion
Acronym: HASA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Klaus Barretto-Lopes (Other)
Responsible Party: Sponsor-Investigator, Klaus Barretto-Lopes, Professor in Orthodontics, Rio de Janeiro State University
Organization: Rio de Janeiro State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HASA
Record Dates: First submitted 2015-03-26; First posted 2015-04-08 (Estimated); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Malocclusion, Angle Class II
Keywords: Orthodontic Appliances, Functional; Herbst Appliance; Malocclusion, Angle Class II
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Orthodontic Appliances, Functional

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Herbst appliance with skeletal anchorage (Experimental): Group treated with the Herbst appliance with indirect skeletal anchorage in mini-implants.
  Interventions: Device: Herbst appliance with skeletal anchorage
- Herbst appliance with dental anchorage (Active Comparator): Group treated with the conventional Herbst appliance with dental anchorage.
  Interventions: Device: Herbst appliance with dental anchorage
- Twin-Block appliances (Active Comparator): Group treated with Twin-Block appliance.
  Interventions: Device: Twin-Block appliance

INTERVENTIONS:
Device: Herbst appliance with skeletal anchorage — Group treated with the Herbst appliance with indirect skeletal anchorage in mini-implants.
  Arms: Herbst appliance with skeletal anchorage
Device: Herbst appliance with dental anchorage — Group treated with the conventional Herbst appliance with dental anchorage.
  Arms: Herbst appliance with dental anchorage
Device: Twin-Block appliance — Group treated with Twin-Block appliance
  Arms: Twin-Block appliances

SUMMARY:
The purpose of this study is to determine if the Herbst appliance with indirect skeletal anchorage in mini-implants is capable of preventing excessive inclination of the lower incisors at the end of the treatment when compared to the Herbst appliance with dental anchorage and Twin-Block appliances in patients with Class II malocclusion and overjet ≥ 6 mm.

DETAILED DESCRIPTION:
2a. Background

The prevalence of the Angle Class II malocclusion is high, comprising almost half of known orthodontic problems (Silva Filho et al., 1990; Proffit et al., 1998). The Class II malocclusion is frequently responsible for negative aesthetic of the facial profile. This can result in psychosocial problems, principally in the Angle Class II, division I malocclusion because of the pronounced projection of the anterior superior teeth. This projection has also been related to fracture and avulsion of the anterior superior teeth.

Different types of appliances had been developed for the treatment of the Angle Class II malocclusion. Among these, functional orthopedic appliances have been used because they can correct Class II malocclusion with better improvement in the growth of the mandible when compared to headgears, which also can correct the problem, but with better restriction of the growth of the maxilla (Tulloch et al., 1997).

The Herbst appliance is a fixed functional orthopedic appliance that is often used because of its non-compliance-nature and the positive results achieved. Emil Herbst created the Herbst appliance in the 1910s (Pancherz; Ruf, 2008), but it was forgotten for decades. Only in the 1970s, Pancherz began a study of the Herbst appliance, and reported the positive results obtained in treatment of the Class II, division I malocclusion (Pancherz, 1979). Several subsequent studies of the Herbst appliance provided new scientific evidence of its benefits.

Nowadays, the Herbst appliance is often used in the treatment of Class II malocclusions, because of its efficiency (Bremen, Pancherz, 2008) and also because of the positive effects in orthodontic and orthopedic correction (Franchi et al., 1999). However, some investigators have stated that the correction of a Class II malocclusion is a result of anchorage loss, and could be responsible for negative effects on the lower incisors such as protrusion and gingival recession (Pancherz, 1979; Pancherz; Hansen, 1986; Pancherz; Hansen, 1988; Schütz et al., 2002; Vigorito; Yared et al., 2006; Dominguez, 2007).

Some attempts have been made to reduce the negative effects on lower incisors caused by the Herbst appliance, such as increasing the number of teeth in the mandibular anchorage, using soft-tissue anchorage, splints, and cast splints anchorage (Weschler et al., 2005; El-Fateh et al., 2011). However, these attempts were unsuccessful.

With the intention of solving these problems, a mini-implant prototype was developed for Herbst appliance anchorage (Barretto-Lopes, 2004). Mini-implants and implants have been used as anchors in orthodontics, for different purposes in different locations (Kanomi, 1997; Deguchi et al., 2003; Miyawaki et al., 2003). Some investigators have suggested the use of mini-implants as orthopedic anchors in animals (Smalley et al., 1988; De Pauw et al., 1999) and in the treatment of Class III malocclusions with retrusive maxillae in humans (Enacar et al., 2003, DeClerck et al., 2010; Heyman et al., 2010). However, there is little information about the use of mini-implants as an orthopedic anchor in the treatment of Class II malocclusions.

Therefore, a first in vitro study was developed to test the flexural resistance of the mini-implant prototypes developed for Herbst appliance anchorage (Barretto-Lopes, 2010, 2010). Subsequently, a question arose with respect to the resistance strength of these mini-implant prototypes when inserted in the bone, and a second ex vivo study was designed to evaluate if the mini-implant prototypes were capable of withstanding orthopedic forces in Minipigs br 1, and to compare the prototype resistance between the sites of insertion. The results showed that the mini-implant prototypes inserted in bone were capable of withstanding orthopedic forces (20.55 kgf for the mandible and 13.86 kgf for the maxilla), and the anterior region of the mandible could withstand statistically significant higher forces than the posterior region of the maxilla (Barretto-Lopes et al., 2012).

The next step was to test the Herbst with skeletal anchorage in humans and a pilot study was performed in patients to test the Herbst appliance with direct anchorage in mini-implants. However, the mini-implants presented mobility in the three cases tested and the trial was suspended.

Probably the direct load in mini-implants would be the reason of the system failure and a second pilot study in humans was carried out using the Herbst appliance with indirect anchorage in mini-implants. This system proved to be stable.

Thus, an in vivo study is necessary to evaluate the effect of the Herbst appliance with indirect anchorage in mini-implants on the lower incisors at the end of treatment compared to the Herbst appliance with dentoalveolar anchorage. Secondarily, this study could evaluate other dental effects and skeletal effects in the maxilla and mandible, resulting from the use of two types of anchoring.

2b. Objectives

Primary objective To determine if the Herbst appliance with indirect skeletal anchorage in mini-implants is capable of preventing excessive inclination of the lower incisors at the end of the treatment when compared to Herbst appliance with dental anchorage and Twin-Block appliances in patients with Class II malocclusion.

Secondary objectives To evaluate the changes occurred on mandible, maxilla, relationship between maxilla and mandible, lower molar and upper molar at the end of the treatment with the Herbst appliance with skeletal and dental anchorage, and Twin-Block appliances in patients with Class II malocclusion.

3-12. Methods

3a. Study design

According to the norms of the CONSORT STATEMENT (Moher et al., 2010), this study will be clinical with intervention, in which the allocation of the subjects will be randomized (block randomization). This study will be parallel, stratified by gender, with blinding for the outcome evaluators. The primary purpose of this study will be treatment.

4b. Participants - Settings and locations where the data are collected

The treatment will be performed in the Orthodontics Clinic of Rio de Janeiro State University. This public university serves a predominantly low-income population located in the Vila Isabel neighborhood in northern Rio de Janeiro State, Brazil. The estimated population size is 81,858 habitants (IBGE - CENSO 2000). Data will be collected from April 2015 through August 2016.

5. Interventions

Three groups will receive treatment. Group 1 will be treated with the Herbst appliance with dental anchorage for 12 months. Group 2 will be treated with the Herbst appliance with skeletal anchorage in mini-implants for 12 months. Group 3 will be treated with Twin-Block appliances.

7a. Sample size

The open source software developed by Harvard University (http://hedwig.mgh.harvard.edu/sample_size/js/js_parallel_quant.html) was used for the sample size calculation. The main outcome measure was the difference between lower incisor proclination before and after treatment. Standard deviation of 1.31 (Martin, Pancherz, 2009) with a two-tailed curve was considered. Difference in means of 2 mm was used as minimal detectable difference. This value was based on a question answered by Professors and Post graduation students who reported a reduction of 2 mm as clinically significant. The significance level will be ≤ 5% and the power of the study will be 80%.

Therefore, 57 subjects will be needed, with 19 subjects in each group. An Intention-to-treat analysis will be performed to deal with dropouts and multiple imputation will be used to deal with missing data. The treatment time will be, approximately, 12 months.

7b. Interim analysis and stopping guidelines

In the group with indirect skeletal anchorage, in case of mobility in the mini-implants in any subject, the load will be removed for about one month. After that, the load will be restored. If the mobility persists, the mini-implant will be removed and reinserted in another site. If mobility occurs again, this subject will be reallocated to the group with dental anchorage. The same procedure will be followed in case of failure of the mini-implant.

8. Randomization

8a. Sequence generation

The randomization of the clinical research will be done with a randomized list, using the first generator from the site www.randomization.com (Pandis et al., 2011).

8b. Type

The type of randomization will be block randomization. In this approach, after the selection of the subjects according to the eligibility criteria, the sample will be separated into 10 blocks with 6 subjects in each.

9. Allocation and concealment mechanism

The sequence of allocation will be concealed in sequential opaque envelopes numbered from 1 to 60, with the treatment modality.

10. Implementation

Before the beginning of the research, the secretary of the Department of Orthodontics of the Faculty of Dentistry of the University of the State of Rio de Janeiro will be responsible for the implementation of the randomization (generation and storage of the randomized list, allocation concealment and treatment assignment). The subjects will write their names on the numbered envelopes, and will open the envelopes to learn the treatment for which they were selected. After that, the envelopes will be closed with the type of treatment selected for storage of the information.

11. Blinding

Blinding will be carried out only for the data analysis because the researchers, participants and subjects will know the treatment modality. Therefore, a person who does not know in which group a subject was treated will analyze the data.

12. Statistical methods

For the primary and secondary outcome measures, the data analysis will be performed using SPSS statistical software package (version 12.0, Chicago). Means, standard deviations, and ranges of the dental and skeletal measures will be calculated for the Herbst appliance with dental anchorage and for the Herbst appliance with indirect skeletal anchorage. Statistical differences will be assessed using analysis of variance. The Wilcoxon's test will be used to assess dental and skeletal differences between the Herbst with dental anchorage and Herbst with indirect skeletal anchorage. Measurements will be repeated after 1 week by an examiner, and intraexaminer correlation coefficients (ICC) will be used to evaluate the reliability of repeated measures. A 1-sample test will be performed on duplicate measurements to test for systematic errors.

ELIGIBILITY:
Inclusion Criteria:

* Teenagers aged from 10 to 14 years old (both genders)
* Parental permission with a signed consent form
* Referral from the Orthodontics Clinic of the State of Rio de Janeiro University or private clinics
* Presenting Class II, Division 1 malocclusion with convex profile and minimum overjet of 6 mm in permanent dentition.

Exclusion Criteria:

* Missing teeth.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Lower incisors position changes as measured by tomographic superimposition of the mandible. | 12 months
  Comparison in lower incisors position between the two groups at the end of the treatment.

SECONDARY OUTCOMES:
Morphological mandible changes as measured by tomographic superimposition of the cranial base. | 12 months
  Comparison between the changes of the mandible in the two groups at the end of the treatment.
Maxilla changes as measured by tomographic superimposition of the cranial base. | 12 months
  Comparison between the changes of the maxilla in the two groups at the end of the treatment.
Changes in relationship between maxilla and mandible as measured by tomographic superimposition of the cranial base. | 12 months
  Comparison between the changes of the relationship between the maxilla and the mandible in the two groups at the end of the treatment.
Lower molar position changes as measured by tomographic superimposition of the mandible. | 12 months
  Comparison between the changes of the lower molar in the three groups at the end of the treatment.
Upper molar position changes as measured by tomographic superimposition of the maxilla. | 12 months
  Comparison between the changes of the upper molar in the three groups at the end of the treatment.
Facial changes as measured by tomographic superimposition of the face | 12 months
  Comparison between the facial changes in the three groups.
Upper airway changes measured by tomographic comparison of spaces of the Nasopharynx (NP), Oropharynx (OP), Hypopharynx (HP) and the end of the Pharynx (P) | 12 months
  Comparison between airway changes between the three groups

CONTACTS AND LOCATIONS:
Overall Officials: Klaus B Lopes, PhD, Principal Investigator — Rio de Janeiro State University; Kevin D O'Brien, PhD, Study Director — University of Manchester; José Augusto M Miguel, PhD, Study Chair — Rio de Janeiro State University; Nathália Palomares, MSc, Study Director — Rio de Janeiro State University
Locations (1):
- Rio de Janeiro State University, Rio de Janeiro, Brazil

REFERENCES:
- [Background] De Pauw GA, Dermaut L, De Bruyn H, Johansson C. Stability of implants as anchorage for orthopedic traction. Angle Orthod. 1999 Oct;69(5):401-7. doi: 10.1043/0003-3219(1999)0692.3.CO;2. PMID 10515136
- [Background] Martin J, Pancherz H. Mandibular incisor position changes in relation to amount of bite jumping during Herbst/multibracket appliance treatment: a radiographic-cephalometric study. Am J Orthod Dentofacial Orthop. 2009 Jul;136(1):44-51. doi: 10.1016/j.ajodo.2007.07.027. PMID 19577147
- [Background] Lopes KB, Dominguez GC, Biasi C, Rossi JL. Flexural strength of mini-implants developed for Herbst appliance skeletal anchorage. A study in Minipigs br1 cadavers. Dental Press J Orthod. 2013 Nov-Dec;18(6):124-9. doi: 10.1590/s2176-94512013000600019. PMID 24351160
- [Background] Allais D, Melsen B. Does labial movement of lower incisors influence the level of the gingival margin? A case-control study of adult orthodontic patients. Eur J Orthod. 2003 Aug;25(4):343-52. doi: 10.1093/ejo/25.4.343. PMID 12938839
- [Background] Artun J, Krogstad O. Periodontal status of mandibular incisors following excessive proclination. A study in adults with surgically treated mandibular prognathism. Am J Orthod Dentofacial Orthop. 1987 Mar;91(3):225-32. doi: 10.1016/0889-5406(87)90450-1. PMID 3469907
- [Background] Deguchi T, Takano-Yamamoto T, Kanomi R, Hartsfield JK Jr, Roberts WE, Garetto LP. The use of small titanium screws for orthodontic anchorage. J Dent Res. 2003 May;82(5):377-81. doi: 10.1177/154405910308200510. PMID 12709505
- [Background] El-Fateh T, Ruf S. Herbst treatment with mandibular cast splints--revisited. Angle Orthod. 2011 Sep;81(5):820-7. doi: 10.2319/101010-591.1. Epub 2011 Mar 28. PMID 21446867
- [Background] Enacar A, Giray B, Pehlivanoglu M, Iplikcioglu H. Facemask therapy with rigid anchorage in a patient with maxillary hypoplasia and severe oligodontia. Am J Orthod Dentofacial Orthop. 2003 May;123(5):571-7. doi: 10.1067/mod.2003.S0889540603000520. PMID 12750679
- [Background] De Clerck H, Cevidanes L, Baccetti T. Dentofacial effects of bone-anchored maxillary protraction: a controlled study of consecutively treated Class III patients. Am J Orthod Dentofacial Orthop. 2010 Nov;138(5):577-81. doi: 10.1016/j.ajodo.2009.10.037. PMID 21055597
- [Background] Franchi L, Baccetti T, McNamara JA Jr. Treatment and posttreatment effects of acrylic splint Herbst appliance therapy. Am J Orthod Dentofacial Orthop. 1999 Apr;115(4):429-38. doi: 10.1016/s0889-5406(99)70264-7. PMID 10194289
- [Background] Hansen K, Koutsonas TG, Pancherz H. Long-term effects of Herbst treatment on the mandibular incisor segment: a cephalometric and biometric investigation. Am J Orthod Dentofacial Orthop. 1997 Jul;112(1):92-103. doi: 10.1016/s0889-5406(97)70279-8. PMID 9228847
- [Background] Heymann GC, Cevidanes L, Cornelis M, De Clerck HJ, Tulloch JF. Three-dimensional analysis of maxillary protraction with intermaxillary elastics to miniplates. Am J Orthod Dentofacial Orthop. 2010 Feb;137(2):274-84. doi: 10.1016/j.ajodo.2009.07.009. PMID 20152686
- [Background] Kanomi R. Mini-implant for orthodontic anchorage. J Clin Orthod. 1997 Nov;31(11):763-7. No abstract available. PMID 9511584
- [Background] Miyawaki S, Koyama I, Inoue M, Mishima K, Sugahara T, Takano-Yamamoto T. Factors associated with the stability of titanium screws placed in the posterior region for orthodontic anchorage. Am J Orthod Dentofacial Orthop. 2003 Oct;124(4):373-8. doi: 10.1016/s0889-5406(03)00565-1. PMID 14560266
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; Consolidated Standards of Reporting Trials Group. CONSORT 2010 Explanation and Elaboration: Updated guidelines for reporting parallel group randomised trials. J Clin Epidemiol. 2010 Aug;63(8):e1-37. doi: 10.1016/j.jclinepi.2010.03.004. Epub 2010 Mar 25. PMID 20346624
- [Background] Pancherz H. The mandibular plane angle in activator treatment. Angle Orthod. 1979 Jan;49(1):11-20. doi: 10.1043/0003-3219(1979)0492.0.CO;2. PMID 283705
- [Background] Pancherz H, Hansen K. Occlusal changes during and after Herbst treatment: a cephalometric investigation. Eur J Orthod. 1986 Nov;8(4):215-28. doi: 10.1093/ejo/8.4.215. No abstract available. PMID 3466794
- [Background] Pancherz H, Hansen K. Mandibular anchorage in Herbst treatment. Eur J Orthod. 1988 May;10(2):149-64. doi: 10.1093/ejo/10.2.149. No abstract available. PMID 3164681
- [Background] Pandis N, Polychronopoulou A, Eliades T. Randomization in clinical trials in orthodontics: its significance in research design and methods to achieve it. Eur J Orthod. 2011 Dec;33(6):684-90. doi: 10.1093/ejo/cjq141. Epub 2011 Feb 14. PMID 21320892
- [Background] Proffit WR, Fields HW Jr, Moray LJ. Prevalence of malocclusion and orthodontic treatment need in the United States: estimates from the NHANES III survey. Int J Adult Orthodon Orthognath Surg. 1998;13(2):97-106. PMID 9743642
- [Background] Ruf S, Hansen K, Pancherz H. Does orthodontic proclination of lower incisors in children and adolescents cause gingival recession? Am J Orthod Dentofacial Orthop. 1998 Jul;114(1):100-6. doi: 10.1016/s0889-5406(98)70244-6. PMID 9674687
- [Background] Smalley WM, Shapiro PA, Hohl TH, Kokich VG, Branemark PI. Osseointegrated titanium implants for maxillofacial protraction in monkeys. Am J Orthod Dentofacial Orthop. 1988 Oct;94(4):285-95. doi: 10.1016/0889-5406(88)90053-4. PMID 3177282
- [Background] Tulloch JF, Phillips C, Koch G, Proffit WR. The effect of early intervention on skeletal pattern in Class II malocclusion: a randomized clinical trial. Am J Orthod Dentofacial Orthop. 1997 Apr;111(4):391-400. doi: 10.1016/s0889-5406(97)80021-2. PMID 9109584
- [Background] Weschler D, Pancherz H. Efficiency of three mandibular anchorage forms in Herbst treatment: a cephalometric investigation. Angle Orthod. 2005 Jan;75(1):23-7. doi: 10.1043/0003-3219(2005)0752.0.CO;2. PMID 15747811
- [Background] Yared KF, Zenobio EG, Pacheco W. Periodontal status of mandibular central incisors after orthodontic proclination in adults. Am J Orthod Dentofacial Orthop. 2006 Jul;130(1):6.e1-8. doi: 10.1016/j.ajodo.2006.01.015. PMID 16849063
- [Derived] Chavez-Sevillano MG, Carvalho FAR, Miguel JAM, Batista KBDSL, Fernandes LQP, Blanco-Victorio DJ, Quintao CCA. Three-dimensional condyle and glenoid fossa alterations after class II treatment with twin block and herbst functional appliances - a randomized clinical trial. Eur J Orthod. 2025 Jun 12;47(4):cjaf038. doi: 10.1093/ejo/cjaf038. PMID 40795311